CLINICAL TRIAL: NCT02899143
Title: Trial of Short-Course Antimicrobial Therapy for Sepsis in Intensive Care
Brief Title: Short-course Antimicrobial Therapy in Sepsis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Santa Maria delle Croci (Other)
Responsible Party: Principal Investigator, Vincenzo De Santis, Medical Doctor, Ospedale Santa Maria delle Croci
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1599
Record Dates: First submitted 2016-09-08; First posted 2016-09-14 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Infection; Sepsis; Severe Sepsis; Septic Shock
MeSH Terms: conditions — Infections; Sepsis; Shock, Septic | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 5-days (Experimental): 5-days targeted antibiotic therapy
  Interventions: Drug: Antibiotic
- Group 10-days (Other): 10-days targeted antibiotic therapy
  Interventions: Drug: Antibiotic

INTERVENTIONS:
Drug: Antibiotic — Targeted antimicrobial therapy

SUMMARY:
The purpose of this study is to compare the effect of a short course antimicrobial therapy (5-days) versus a 10-days therapy on sepsis-related organ dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received antibiotics for presumed infection

Exclusion Criteria:

* Prolonged therapy (eg, endocarditis)
* Severe immunosuppression
* Severe infections (due to viruses, parasites, or Mycobacterium tuberculosis)
* Patients previously infected or colonized with multidrug resistant pathogens and moribund patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2016-09; Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
sepsis-related organ dysfunction | 14-days
  Score used to track a person's status during the stay in an intensive care unit (ICU) to determine the extent of a person's organ function or rate of failure. The Sequential Organ Failure Assessment (SOFA) score numerically quantifies the number and severity of failed organs. Higher values represent worse outcome. A score of 0 is given for normal function through to 4 for most abnormal. The systems studied are: respiratory, coagulation, hepatic, cardiovascular, central nervous system, and renal.

SECONDARY OUTCOMES:
Hospital mortality | 30-days
  In hospital mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo De Santis, Principal Investigator — Ospedale Santa Maria Delle Croci, Ravenna, AUSL Romagna
Locations (4):
- Italy (4):
  - Ospedale Umberto I, Lugo, Ravenna
  - Azienda Ospedaliera S.Croce e Carle - Ospedale S.Croce, Cuneo
  - ASST Fatebenefratelli Sacco, Milan
  - Ospedale Santa Maria Delle Croci, Ravenna